CLINICAL TRIAL: NCT01491477
Title: Study of Recombinant Human Bone Morphogenetic Protein-2 and Absorbable Collagen Sponge With the Cornerstone-SR™ Allograft Ring and the ATLANTIS™ Anterior Cervical Plate System in Treatment of Patients With Degenerative Cervical Disc Disease
Brief Title: INFUSE ® Bone Graft/CORNERSTONE-SR® Allograft Ring/ATLANTIS® Anterior Cervical Plate System Pivotal Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01-04
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2011-12

CONDITIONS: Degenerative Cervical Disc Disease
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INFUSE™ Bone Graft (Experimental)
  Interventions: Device: INFUSE™ Bone Graft/CORNERSTONE-SR™ /ATLANTIS™
- Autogenous bone (Active Comparator)
  Interventions: Device: Autogenous bone/CORNERSTONE-SR™ /ATLANTIS™

INTERVENTIONS:
Device: INFUSE™ Bone Graft/CORNERSTONE-SR™ /ATLANTIS™ — Cornerstone-SR™ allograft bone containing recombinant human Bone Morphogenetic Protein (rhBMP-2) soaked into an absorbable collagen sponge (ACS) used in conjunction with ATLANTIS™ anterior cervical plate system.
  Other Names: Recombinant human bone morphogenetic protein-2
  Arms: INFUSE™ Bone Graft
Device: Autogenous bone/CORNERSTONE-SR™ /ATLANTIS™ — Cornerstone-SR™ allograft bone packed with autogenous iliac crest bone graft used in conjunction with ATLANTIS™ anterior cervical plate system.
  Other Names: Autograft
  Arms: Autogenous bone

SUMMARY:
The purpose of this trial is to evaluate the implant (INFUSE™ BONE GRAFT/CORNERSTONE-SR™ Allograft Ring/ATLANTIS™ Anterior Cervical Plate system) as a method of facilitating spinal fusion in patients with cervical symptomatic degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical disc disease defined as: intractable radiculopathy and/or myelopathy with at least one of the following items producing symptomatic nerve root and/or spinal cord compression which is documented by diagnostic imaging procedures:

   * herniated disc;
   * osteophyte formation;
   * decreased disc height;
   * thickening of ligamentous tissue;
   * disc degeneration; and/or
   * facet joint degeneration.
2. Has preoperative Neck Disability Index score > 30;
3. Has single cervical disc disease level requiring fusion from C2 to C7;
4. No previous surgical intervention at the involved fusion level;
5. Unresponsive to nonoperative treatment for approximately six weeks or has the presence of progressive symptoms or signs of nerve root or spinal cord compression in face of continued nonoperative management;
6. Is at least 18 years of age, inclusive at time of surgery;
7. If of child-bearing potential, patient is non-pregnant, non-nursing, and agrees to use adequate contraception for 1 year following surgery;
8. Is willing and able to comply with study plan and sign the consent form.

Exclusion Criteria:

1. Has cervical spinal condition requiring surgical treatment other than symptomatic cervical disc disease at the involved level.
2. Has a condition which requires postoperative medications that interfere with fusion, such as steroids or prolonged non-steroidal anti-inflammatory drugs excluding routine perioperative anti-inflammatory drugs. This does not include low dose aspirin for prophylactic anticoagulation.
3. Has been previously diagnosed with osteopenia, or osteomalacia.
4. Has any of the following that may be associated with a diagnosis of osteoporosis (if "Yes" to any of the below risk factors, a DEXA Scan will be required to determine eligibility).

   1. Postmenopausal Non-Black female over 60 years of age and weighs less than 140 pounds.
   2. Postmenopausal female that has sustained a non-traumatic hip, spine, or wrist fracture.
   3. Male over the age of 70.
   4. Male over the age of 60 that has sustained a non-traumatic hip or spine fracture.

   If the level of BMD is a T score of -3.5 or a T score of -2.5 with vertebral crush fracture, the patient is excluded from the study.
5. Has presence of active malignancy or prior history of malignancy, except for basal cell carcinoma of the skin.
6. Has overt or active bacterial infection, either local or systemic.
7. Has a documented titanium alloy allergy or intolerance.
8. Is mentally incompetent. If questionable, obtain psychiatric consult.
9. Is a prisoner.
10. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug usage.
11. Has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., steroids or methotrexate), excluding routine perioperative anti-inflammatory drugs.
12. Has a history of autoimmune disease (Systemic Lupus Erythematosus or Dermatomyositis).
13. Has a history of exposure to injectable collagen implants.
14. Has a history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
15. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/ACS implantation.
16. Has received any previous exposure to any/all BMP's of either human or animal extraction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2002-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Overall Success | 12 month
  A patient will be considered an overall success if all of the following conditions are met:
  1. fusion;
  2. pain/disability (Neck Disability Index) Improvement;
  3. maintenance or improvement in neurological status;
  4. no serious adverse event classified as "implant associated" or "implant/surgical procedure associated";
  5. no additional surgical procedure classified as a "failure".

SECONDARY OUTCOMES:
Disc Height Measurement | 12 month
General Health Status (SF-36) | 12 month
Pain Status (neck pain, arm pain) | 12 month
Patient Satisfaction | 12 month
Patient Global Perceived Effect | 12 month